CLINICAL TRIAL: NCT02058446
Title: An Open-label, Postmarketing Study of Amlodipine/Valsartan Single-Pill Combination for the Treatment of Hypertension
Brief Title: PMS Study of Amlodipine/Valsartan for the Treatment of Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSHAM1301
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2014-02

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): Amlodipine/Valsartan Single-Pill Combination
  Interventions: Drug: Amlodipine/Valsartan

INTERVENTIONS:
Drug: Amlodipine/Valsartan — Amlodipine/Valsartan: 5 mg/80 mg
  Other Names: Am-Daiwen®

SUMMARY:
The antihypertensive effect of Amlodipine/Valsartan combination has been evaluated in worldwide populations including Asian patients. The study primarily aims to evaluate the effectiveness of Amlodipine/Valsartan combination in patients with essential hypertension in Taiwan using a prospective, open-label, non-randomized approach.

The study also wants to investigate the safety of Amlodipine/Valsartan combination during the 6-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 20-80 years of age
* Patients with essential hypertension (90 mmHg ≤ DBP ≤ 110 mmHg and/or 140 mmHg ≤ SBP ≤ 180 mmHg) whose BP is not adequately controlled with amlodipine (or another CCB) alone or with valsartan (or another ARB) alone, or with any antihypertensive monotherapy.
* Agree to and are able to follow the study procedures
* Understand the nature of the study, and have signed informed consent forms

Exclusion Criteria:

* Patients with any of the following conditions:

  1. Malignant (or history of malignant) hypertension
  2. Secondary hypertension
  3. Severe hypertension (mean sitting DBP ≥ 110 mmHg and/or mean sitting SBP ≥ 180 mmHg)
  4. A history of hypertensive encephalopathy or cerebrovascular accident
  5. Cerebrovascular accident, myocardial infraction within 3 months, or any type of revascularization
  6. New York Heart Association class III -IV congestive heart failure
  7. Second- or third-degree heart block
  8. Angina pectoris
  9. Significant arrhythmia or valvular heart disease
  10. Significant pancreatic, hepatic, or renal disease
  11. Diabetes requiring insulin treatment or poorly controlled type 2 diabetes
* Patients with known contraindication or a history of allergy to CCBs or ARBs.
* Female patients who are pregnant or lactating.
* Male or female patients of child-bearing potential who do not agree to use an effective method of contraception during the study
* Patients is currently participating in any other clinical trial within 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the change from baseline in office SBP measurements by cuff assessments at the end of the 6-week study period. | 6 weeks from baseline

SECONDARY OUTCOMES:
To evaluate the change from baseline in office DBP measurements by cuff assessments after 6 weeks of treatment | 6 weeks from baseline
To evaluate the percentage of subjects who achieve BP goal as measured by cuff assessments (<140/90 mmHg) after 6 weeks of treatment | 6 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Yang Wang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan